CLINICAL TRIAL: NCT04654520
Title: A Randomized Study of Primary Tumor Radiotherapy Omitting Clinical Target Volume for Patients With Stage Ⅳ NSCLC
Brief Title: A Randomized Study of Primary Tumor Radiotherapy for Patients With Stage Ⅳ NSCLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guizhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ⅳ-NSCLC-OCTV
Record Dates: First submitted 2020-11-29; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Radiotherapy; Nonsmall Cell Lung Cancer, Stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug therapy combined with radiotherapy for primary tumor omitted CTV (Experimental): * IMRT (omitted CTV) concurrent with systemic chemotherapy on paticipants of kown negative gene mutation .After it, the paticipants may choose immunotherapy.
  * IMRT (omitted CTV) concurrent with targeted drug on paticipants of kown sensitive gene mutation.
  Interventions: Other: Drug therapy concurrent radiotherapy for primary tumor omitted CTV
- Drug therapy combined with radiotherapy for primary tumor with CTV (No Intervention): * IMRT (with CTV) concurrent with systemic chemotherapy on paticipants of kown negative gene mutation .After it, the paticipants may choose immunotherapy.
  * IMRT ((with CTV) concurrent with targeted drug on paticipants of kown sensitive gene mutation.

INTERVENTIONS:
Other: Drug therapy concurrent radiotherapy for primary tumor omitted CTV — Thoracic intensity modulated radiotherapy for primary tumor omitted CTV+Chemotherapy or Targeted drug therapy
  Arms: Drug therapy combined with radiotherapy for primary tumor omitted CTV

SUMMARY:
The aim of this randomized study is to investigate local tumor control, survival outcomes,and complications on patients of stage Ⅳ non small-cell lung cancer ,whom based on medication with concurrent primary radiotherapy omitting clinical tumor volume.

DETAILED DESCRIPTION:
Cancer Statistics,（2020）states that low lung cancer survival rates reflect the large proportion of patients (57%) diagnosed with metastatic disease, for which the 5-year relative survival rate is 5%.With the development of three-dimensional radiotherapy technology, the wide application of comprehensive treatment concept, and the understanding of the relationship between different metastatic state and survival of stage IV NSCLC, prospective and retrospective studies have confirmed that systemic therapy combined with primary tumor three-dimensional radiation Treatment is more conducive to improving symptoms and prolonging survival than medication alone. Some retrospective analysises of stage III NSCLC, omitting clinical target volume of primary tumor with intensity modulated radiotherapy showed no reduction in local control rate and survival time.Omitted CTV in Ⅳ NSCLC patients with primary tumor radiotherapy can make smaller target area, which could push up most of the local stage of late Ⅳ NSCLC patients with primary tumor radiation dose. Prospective studies are needed to further clarify whether omission of target areas may affect local control time, survival time, and radioactive toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathological or cytological diagnosis, stage IV [UICC 2017 staging eighth edition] NSCLC patients;
* initial treatment (previously did not receive any treatment), it is recommended to complete the detection of driver genes (EGFR / ALK / ROS1) (tissue, blood);
* Age 18 to 80 years old, physical status score ECOG 0 to 2 or KPS ≥ 70 (see Annex 2); Metastatic lesions in the distant area: conscious when brain metastasis; the number of metastatic lesions in the lung does not affect lung function and may be treated with primary and/or partial metastases;
* no radiotherapy, targeted drug therapy and chemotherapy contraindications;
* primary tumor radiotherapy requires IMRT technology;
* Plan the design to give the primary tumor prescription dose (DTGTV) under the damage control threshold criteria;
* The planned dose includes 100% GTV, 90% of the prescribed dose includes 98%~100% of PTV [planned target dose (DTPTV)]; normal lung (full lung volume minus GTV volume) V20 ≤ 32%, MLD≤20Gy;
* metastatic tumor radiotherapy is a three-dimensional radiotherapy technique (IMRT/SRT/SBRT/VMAT, etc.), and large-segment radiotherapy.
* Subjects have no major organ dysfunction, or laboratory test indicators must meet the following requirements: Hematology: normal range according to laboratory standards; cardiac function: normal range; liver function: normal range; renal function: normal range Lung function: FEV1>50%, impaired light-moderate lung function.
* Informed consent (radiation, medication) before treatment;
* The patient has good compliance with the treatment and follow-up received.

Exclusion Criteria:

* Patients who do not meet the pathological type, stage, and survival status of the inclusion criteria;
* patients with malignant pericardial effusion; Diffuse liver metastasis, intrapulmonary metastasis and has seriously affected patients with liver and lung function;
* Patients with uncontrolled hypertension, diabetes, unstable angina, history of myocardial infarction, or symptomatic congestive heart failure or uncontrolled arrhythmias in the past 12 months; clinically diagnosed heart valve disease;
* Active period of disease caused by bacteria, fungi or viruses; mental disorders; impaired severe lung function;
* pregnant, lactating patients;
* Patients with a history of other active malignancies other than small cell lung cancer before entering the group; non-melanoma skin basal cell carcinoma, in situ cervical cancer, and cured early prostate cancer;
* Patients with allergies and no known alternatives to known or suspected drugs in any study;
* Patients with poor compliance;
* Researchers believe that it is not appropriate to participate in this test.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2020-12-15 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Local regional progression-free survival（LRPFS） | Up to 5 years
  LRPFS is defined as the duration of time from start of treatment to time of progression or recurrence, whichever occurs first.The target lesions is only for primary tumor and regional positive lymph nodes.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 5 years
  Overall survival is defined as the time interval from date of diagnosis to date of death from any cause.
Progression-free survival (PFS) | Up to 5 years
  PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
Adverse events (toxicities) | Up to 5 years
  The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Bing Lu, Bachelor, Principal Investigator — Affiliated Hospital of Guizhou Medical University
Locations (1):
- Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou, China

IPD SHARING:
Plan to Share IPD: No